CLINICAL TRIAL: NCT05657808
Title: Radicle™ Rest 2: A Randomized, Blinded, Placebo-Controlled Direct-to-Consumer Study of Health and Wellness Products on Sleep and Other Health Outcomes
Brief Title: Radicle Rest 2: A Study of Health and Wellness Products on Sleep and Health Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radicle Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: RADX-2301
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Sleep; Sleep Disturbance; Sleep Disorder
MeSH Terms: conditions — Parasomnias; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on sex at birth then randomized to one of the study arms
Who Masked: Participant, Investigator
Masking Description: The investigator is blinded to the participants' study product assignment. Participants are blinded to the study product they are assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Placebo Control 1 (Placebo Comparator): Rest Product Form 1 - control
  Interventions: Dietary Supplement: Placebo Control Form 1
- Placebo Control 2 (Placebo Comparator): Rest Product Form 2 - control
  Interventions: Dietary Supplement: Placebo Control Form 2
- Active Product 1.1 (Experimental): Rest Product Form 1 - active product 1
  Interventions: Dietary Supplement: Rest Study Active Product 1.1 Usage
- Active Product 1.2 (Experimental): Rest Product Form 1 - active product 2
  Interventions: Dietary Supplement: Rest Study Active Product 1.2 Usage
- Active Product 2.1 (Experimental): Rest Product Form 2 - active product 1
  Interventions: Dietary Supplement: Rest Study Active Product 2.1 Usage
- Active Product 2.2 (Experimental): Rest Product Form 2 - active product 2
  Interventions: Dietary Supplement: Rest Study Active Product 2.2 Usage
- Placebo Control 3 (Placebo Comparator): Rest Product Form 3 - control
  Interventions: Dietary Supplement: Placebo Control Form 3
- Active Product 3.1 (Experimental): Rest Product Form 3 - active product 1
  Interventions: Dietary Supplement: Rest Study Active Product 3.1 Usage
- Placebo Control 4 (Placebo Comparator): Rest Product Form 4 - control
  Interventions: Dietary Supplement: Placebo Control Form 4
- Active Product 4.1 (Experimental): Rest Product Form 4 - active product 1
  Interventions: Dietary Supplement: Rest Study Active Product 4.1 Usage
- Active Product 4.2 (Experimental): Rest Product Form 4 - active product 2
  Interventions: Dietary Supplement: Rest Study Active Product 4.2 Usage
- Active Product 4.3 (Experimental): Rest Product Form 4 - active product 3
  Interventions: Dietary Supplement: Rest Study Active Product 4.3 Usage

INTERVENTIONS:
Dietary Supplement: Rest Study Active Product 1.1 Usage — Participants will use Radicle Rest Active Product 1.1 as directed for a period of 6 weeks.
  Arms: Active Product 1.1
Dietary Supplement: Rest Study Active Product 1.2 Usage — Participants will use Radicle Rest Active Product 1.2 as directed for a period of 6 weeks.
  Arms: Active Product 1.2
Dietary Supplement: Rest Study Active Product 2.1 Usage — Participants will use Radicle Rest Active Product 2.1 as directed for a period of 6 weeks.
  Arms: Active Product 2.1
Dietary Supplement: Rest Study Active Product 2.2 Usage — Participants will use Radicle Rest Active Product 2.2 as directed for a period of 6 weeks.
  Arms: Active Product 2.2
Dietary Supplement: Placebo Control Form 1 — Participants will use Placebo Control Form 1 as directed for a period of 6 weeks.
  Arms: Placebo Control 1
Dietary Supplement: Placebo Control Form 2 — Participants will use Placebo Control Form 2 as directed for a period of 6 weeks.
  Arms: Placebo Control 2
Dietary Supplement: Placebo Control Form 3 — Participants will use Placebo Control Form 3 as directed for a period of 6 weeks.
  Arms: Placebo Control 3
Dietary Supplement: Rest Study Active Product 3.1 Usage — Participants will use Radicle Rest Active Product 3.1 as directed for a period of 6 weeks.
  Arms: Active Product 3.1
Dietary Supplement: Placebo Control Form 4 — Participants will use Placebo Control Form 4 as directed for a period of 6 weeks.
  Arms: Placebo Control 4
Dietary Supplement: Rest Study Active Product 4.1 Usage — Participants will use Radicle Rest Active Product 4.1 as directed for a period of 6 weeks.
  Arms: Active Product 4.1
Dietary Supplement: Rest Study Active Product 4.2 Usage — Participants will use Radicle Rest Active Product 4.2 as directed for a period of 6 weeks.
  Arms: Active Product 4.2
Dietary Supplement: Rest Study Active Product 4.3 Usage — Participants will use Radicle Rest Active Product 4.3 as directed for a period of 6 weeks.
  Arms: Active Product 4.3

SUMMARY:
A randomized, blinded, placebo-controlled direct-to-consumer study assessing the impact of health and wellness products on sleep and other health outcomes.

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled study conducted with adult participants, age 21 and older and residing in the United States.

Eligible participants will (1) endorse a desire for improved sleep, (2) indicate an interest in taking a health and wellness product to potentially help their sleep, and (3) express acceptance in taking a product and not knowing its formulation until the end of the study.

Participants with known liver or kidney disease, heavy drinkers, and those who report they are pregnant, trying to become pregnant, or breastfeeding will be excluded. Those taking certain medications will be excluded.

Self-reported data are collected electronically from eligible participants over 7 weeks. Participant reports of health indicators will be collected during baseline, throughout the active period of study product use, and in a final survey. All study assessments will be electronic; there are no in-person visits or assessments for this real-world evidence study.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 21 years of age and older at the time of electronic consent, inclusive of all ethnicities, races, genders and/or gender identities
* Resides in the United States
* Endorses better sleep as a primary desire
* Selects sleep, looking to improve their sleep, and/or reduce reliance on medications as a reason for their interest in taking a health and wellness product
* Expresses a willingness to take a study product and not know the product identity (active or placebo) until the end of the study

Exclusion Criteria:

* Reports being pregnant, trying to become pregnant, or breastfeeding
* Unable to provide a valid US shipping address
* The calculated validated health survey (PRO) measurement result is less than mild severity/impairment
* Reports a diagnosis of liver or kidney disease
* Reports being a heavy drinker (defined as drinking 3 or more alcoholic beverages per day)
* Unable to read and understand English
* Reports current enrollment in a clinical trial
* Lack of reliable daily access to the internet
* Reports current or recent (within 3 months) use of chemotherapy, immunotherapy, or oral anti-infectives (antibiotics, antifungals, antivirals) to treat an acute infection
* Reports taking medications with a known moderate or severe interaction with any of the active ingredients studied: anticoagulants, a medication that warns against grapefruit consumption, corticosteroids at doses greater than 5 mgs per day, or monoamine oxidase inhibitors (MAOIs)
* Reports a diagnosis of heart disease when a known contraindication exists for any of the active ingredients studied: New York Heart Association (NYHA) Class III or IV congestive heart failure, Atrial fibrillation, Uncontrolled arrhythmias

Ages: 21 Years to 105 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4152 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Change in sleep disturbance | 6 weeks
  Mean difference in sleep disturbance score as assessed by Patient Reported Outcome Measurement System (PROMIS) Sleep Disturbance Short Form 8A (scale 8-40; where higher scores correspond to greater sleep disturbance)

SECONDARY OUTCOMES:
Change in fatigue | 6 weeks
  Mean difference in fatigue score as assessed by PROMIS Fatigue 4A (scale 4-20; where higher scores correspond to more severe fatigue)
Change in cognitive function | 6 weeks
  Mean difference in cognitive function score as assessed by PROMIS Cognitive Function 4A (scale 4-20; where higher scores correspond to greater cognitive function)
Change in anxiety | 6 weeks
  Mean difference in anxiety score as assessed by PROMIS Anxiety 4A (scale 4-20; with higher scores corresponding to more severe anxiety)
Change in mood (emotional distress) | 6 weeks
  Mean difference in mood score as assessed by PROMIS Depression 4A (scale 4-20; where higher scores correspond to more severe depression)
Change in libido | 6 weeks
  Mean difference in libido score as assessed by PROMIS Sexual Interest 2.0 (scale 2-10; where higher scores correspond to greater sexual interest)
Minimal clinical importance difference (MCID) in sleep disturbance | 6 weeks
  Likelihood of achieving a MCID in sleep disturbance, as measured by PROMIS Sleep Disturbance Short Form 8A (scale 8-40; where higher scores correspond to greater sleep disturbance)

CONTACTS AND LOCATIONS:
Overall Officials: Emily K. Pauli, PharmD, Principal Investigator — Radicle Science Inc.
Locations (1):
- Radicle Science, Inc, Del Mar, California, United States

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with researchers outside of Radicle Collaborators on this study.

REFERENCES:
- See also: Radicle Science, Inc — http://radiclescience.com